CLINICAL TRIAL: NCT06080217
Title: Radiofrequency as the New Opportunity in Treating Overactive Bladder and Urgent Urinary Incontinence - a Prospective Randomized Placebo Controlled Study
Brief Title: RF in the Treatment OAB in UUI- a Prospective Randomized Placebo Controlled Study
Acronym: RFandOAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ginekologija Dr. Franić, D.O.O. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ginek dr franic
Record Dates: First submitted 2023-06-22; First posted 2023-10-12 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-06

CONDITIONS: Overactive Bladder Syndrome; Urge Incontinence
Keywords: radiofrequency-overactive bladder-urge incontinence
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): The patients were lying in the lithotomy position with the streTched lower extremities. Probes are placed on the lower part of the abdomen in the area of the bladder (active probe) and on the lumbar spine (passive probe). A capacitive probe in the "free treatment" / "power control" program was used, where high frequency electricity was released to the bladder for 20 minutes with a frequency of 1.0 MHz and energy to maximum 410 C. Initialy, maximum energy of 75% and a frequency of 0.8 MHz was applied, which was reduced depending on the heat that was pleasant for the patient. Then, the power was reduced to 50% and increased the frequency to 1.0 MHz, which also meant moderate energy absorption. The procedure with this energy was continued until the end, and the patients absorbed 18-19 kJ of energy in average.
  Interventions: Device: study group
- placebo group (Sham Comparator): The patients were lying in the lithotomy position with the streched lower extremities. Probes are placed on the lower part of the abdomen in the area of the bladder (active probe) and on the lumbar spine (passive probe) . A capacitive probe in the "free treatment" / "power control" program was used, with NO electricity was released to the bladder for 20 minutes
  Interventions: Device: study group; Device: placebo (sham control)

INTERVENTIONS:
Device: study group — The patients were lying in the lithotomy position with the stretched lower extremities. Probes are placed on the lower part of the abdomen in the area of the bladder (active probe) and on the lumbar spine (passive probe). A capacitive probe in the "free treatment" / "power control" program was used, where high frequency electricity was released to the bladder for 20 minutes with a frequency of 1.0 MHz and energy to maximum 410 C. Initialy, maximum energy of 75% and a frequency of 0.8 MHz was applied, which was reduced depending on the heat that was pleasant for the patient. Then, the power was reduced to 50% and increased the frequency to 1.0 MHz, which also meant moderate energy absorption. The procedure with this energy was continued until the end, and the patients absorbed 18-19 kJ of energy in average.
  Other Names: Capenergy C100 (ref. 533001) with upgrade to C500 (ref. 533005)
Device: placebo (sham control) — The patients were lying in the lithotomy position with the stretched lower extremities. Probes are placed on the lower part of the abdomen in the area of the bladder (active probe) and on the lumbar spine (passive probe). A capacitive probe in the "free treatment" / "power control" program was used, but without any energy transferred through the probe,
  Other Names: Capenergy C100 (ref. 533001) with upgrade to C500 (ref. 533005)
  Arms: placebo group

SUMMARY:
Until now, OAB with or without UUI has been treated mainly in two ways: with behavioral methods and/or patient education or using antimuscarinic drugs and/or beta 3 adrenergic receptor agonists. Unfortunately, the drugs might cause side effects in some women or were insufficiently effective, so the patients abandoned them.

Methods In prospective, randomized, placebo controlled study, 80 women were enrolled, using radiofrequency in treating OAB and UUI. Based on ICIQ-OAB, ICIQ-OAB QoL, and ICIQ-FLUTSsex questionnaires, severity of OAB symptoms, QoL and detailed evaluation of female sexual matters associated with their lower urinary tract symptoms. RF was applied 4 times for 20 minutes, once a week. Two week after the completion of the treatment,as well as 3, 6 and 12 months, the level of OAB and UUI was reassessed and processed it statistically and evaluated the treatment effect.

DETAILED DESCRIPTION:
Criteria for inclusion in the study Women who have clear signs of OAB was included in the study. Also, those women who did not use drugs for the treatment of OAB (antimuscarinics/beta-3 agonists), were included.

Those women who have taken drugs for the treatment of OAB in the past, but stopped (side effects, ineffectiveness) and at least 3 months have passed since the last treatment, were also included in the study.

Exclusion criteria from the study Inserted heart pacemaker, unexplained bleeding from the vagina, inflammation of the vagina and/or uterus or uterine appendages. Bacterial or viral infection, impaired immune system, sclerodermia, radiation treatment, burns in the treatment area. Women with stress urinary incontinence (SUI) or mixed urinary incontinence were not included in the study.

Radiofrequency in the treatment of urinary incontinence

In the study, the radiofrequency device Capenergy model C 100 with an upgrade to the urogynecological model C 500, was used. This device has a 1-channel capacitive and resistive probe for individual use. The mechanism of action is electrotherapy with the help of high-frequency electricity (TECAR).

The use of electromagnetic energy in the organism causes biological and physiological reactions. Since the organism is a conductor of the second level, it consists of a large amount of water with an infinite amount of ions dissolved in it. The application of electromagnetic energy to the organism means the acceleration of metabolic responses at various levels, which are used for therapeutic purposes. TECAR evolution generates energy from 0.8-1.2 MHz that was used for the treatment. Nevertheless, the mechanism of action includes the use of high-frequency electricity of heat gain in the body tissues, as a result of the resistance those tissues offer to the current flowing.

The patients were lying in the lithotomy position with the streched lower extremities. Probes are placed on the lower part of the abdomen in the area of the bladder (active probe) and on the lumbar spine (passive probe) Figure 1. A capacitive probe in the "free treatment" / "power control" program was used, where high frequency electricity was released to the bladder for 20 minutes with a frequency of 1.0 MHz and energy to maximum 410 C. Initialy, maximum energy of 75% and a frequency of 0.8 MHz was applied, which was reduced depending on the heat that was pleasant for the patient. Then, the power was reduced to 50% and increased the frequency to 1.0 MHz, which also meant moderate energy absorption. The procedure with this energy was continued until the end, and the patients absorbed 18-19 kJ of energy in avarage.

Such energy desensitizes the bladder and therefore increases its capacity, increases blood flow and reduces the formation of free radicals , which all together improves the symptoms of OAB and UUI.

ELIGIBILITY:
Inclusion Criteria:

* clear signs of OAB
* did not use drugs for the treatment of OAB (antimuscarinics/beta-3 agonists)
* women who have taken drugs for the treatment of OAB in the past, but stopped at least 3 months prior the entering the study.

Exclusion Criteria:

* Inserted heart pacemaker,
* unexplained bleeding from the vagina,
* inflammation of the vagina and/or uterus or uterine appendages.
* Bacterial or viral infection,
* weakened immune system,
* sclerodermia,
* radiation treatment,
* burns in the treatment area,
* stress urinary incontinence (SUI) or mixed urinary incontinence

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
changed symptoms specific for OAB | 2 weeks, 3 months, 6 months, 12 months
  frequency of urination, nocturia, urgency, incontinence

CONTACTS AND LOCATIONS:
Overall Officials: damir franić, MD PhD, Principal Investigator — Ginekologija Dr. Franić, D.O.O.
Locations (2):
- Slovenia (2):
  - Damir Franić, Rogaška Slatina
  - Outpatient Clinic Ob&Gyn, Rogaška Slatina

IPD SHARING:
Plan to Share IPD: Yes
publication in the peer-review journal
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after completed the study together with 12 months follow-up
Access Criteria: e-mail adress: damir.franic@guest.arnes.si; ginekologija.drfranic@siol.net
URL: http://ginekologija.si